CLINICAL TRIAL: NCT05562960
Title: Plasmapheresis in Amyotrophic Lateral Sclerosis With Autoantibody Against NRIP
Acronym: PALATIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202202042DINC
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Amyotrophic Lateral Sclerosis; Plasmapheresis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALS patients receiving plasmapheresis (Other): Plasmapheresis in ALS patients with different titers of autoantibody against NRIP
  Interventions: Procedure: Plasmapheresis

INTERVENTIONS:
Procedure: Plasmapheresis — Regular plasmapheresis to remove anti-NRIP autoantibody

SUMMARY:
Patient with amyotrophic lateral sclerosis (ALS) having anti-NRIP autoantibody showed titer-dependent detrimental Effects. Plasmapheresis might benefit this subgroup of patients via removal of anti-NRIP autoantibody

ELIGIBILITY:
Inclusion Criteria:

1. Patients with amyotrophic lateral sclerosis (ALS) at the age more than 20 years and having plasma anti-NRIP autoantibody.
2. Agree to receive plasmapheresis intervention.
3. Agree to participate in the trial and receive serial examinations and follow up.

Exclusion Criteria:

1. Patients without plasma anti-NRIP autoantibody.
2. Patients requiring permanent ventilator support for ALS progression.
3. Not able to receive plasmapheresis or trial-related examinations.
4. Under pregnancy.
5. Blood fibrinogen level less than 50 mg/dl.
6. Specific ALS subtypes, including primary lateral sclerosis, progressive muscular atrophy, flail arm syndrome, or flail leg syndrome.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in ALSFRS-R decline | Before (3-month) and after (3-month) intervention
  Change in ALSFRS-R decline before (3-month) and after (3-month) intervention. <ALSFRS-R indicates revised ALS functional rating scale, ranged from 0 to 48 with the higher, the better motor function>

SECONDARY OUTCOMES:
Change in ALSFRS-R decline | Before (3-month) and after (6-month) intervention
  Change in ALSFRS-R decline before (3-month) and after (6-month) intervention
Changes in ALSFRS-R score | Day 0 to days 30, 90, and 180
  Changes in ALSFRS-R score from day 0 to days 30, 90, and 180
Change in force vital capacity | Before intervention and on day 90
  Change in force vital capacity before intervention and on day 90
Change in compound motor action potentials | Before intervention and on day 90
  Change in compound motor action potentials before intervention and on day 90
Changes in anti-NRIP titer | Day 0 to days 30, 90, and 180
  Changes in anti-NRIP titer from day 0 to days 30, 90, and 180
Any adverse effect under plasmapheresis | Within 6 months during and after plasmapheresis
  Any adverse effect during and within 6 months after plasmapheresis

CONTACTS AND LOCATIONS:
Overall Officials: Li-Kai Tsai, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No